CLINICAL TRIAL: NCT04142060
Title: Targeting the PAM50 Her2-Enriched Phenotype With Enzalutamide in Hormone Receptor-Positive/Her2-Negative Metastatic Breast Cancer
Brief Title: Targeting the PAM50 Her2-Enriched Phenotype With Enzalutamide in Hormone Receptor-Positive/Her2-Negative Metastatic BC
Acronym: ARIANNA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of effectiveness
Sponsor: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARIANNA (SOLTI-1502); 2019-002806-28 (EudraCT Number)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: an exploratory, open-label, non-randomized, two-cohort, multicenter, prospective, phase II study which evaluates the effect of enzalutamide on proliferation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): Patients will be dispensed with oral enzalutamide 160 mg (four 40 mg capsules) as a self-administered single oral daily dose, continuously
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Patients will be dispensed with oral enzalutamide 160 mg (four 40 mg capsules) as a self-administered single oral daily dose, continuously.
  Other Names: Xtandi

SUMMARY:
The main hypothesis of the study is that enzalutamide induces a significant proliferative arrest in HR+/HER2-negative breast cancer falling into the PAM50 HER2-E subtype. Currently, enzalutamide clinical development is ongoing in different prostate cancer indications but the breast cancer development program has been discontinued. As the role of the AR in HR-positive breast cancer and the predictive value of previously identified biomarker are still unclear, further research is needed to effectively utilize enzalutamide in this disease.

DETAILED DESCRIPTION:
A strong rationale accumulated over the years suggests that within HR+/HER2-negative breast cancer, tumors falling into the PAM50 HER2-enriched subtype have androgen receptor (AR)-dependency. To test this hypothesis directly in patients' tumors, we propose an exploratory, open-label, non-randomized, two-cohort, multicenter, prospective, phase II study which evaluates the effect of enzalutamide on proliferation after 2 weeks (14-21 days) of treatment in patients with endocrine-resistant, locally advanced or metastatic HR+/HER2-negative breast cancer. After 2 weeks (14-21 days) of treatment, patients will continue enzalutamide. Exemestane will be allowed to be added to enzalutamide per investigator discretion and will be administered until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
* Subjects with progression on or following at least 1 prior standard of care systemic anti-cancer therapy.
* Female and male patients.
* Performance status of 0-2.
* Age ≥18 years.
* Pre/peri-menopausal and post-menopausal women are allowed; menopausal status is relevant for the requirement of goserelin, triptorelin or leuprolide to be used concomitantly with enzalutamide. Post-menopausal status is defined either by:

  * Prior bilateral oophorectomy or
  * Age ≥60 or
  * Age < 60 and amenorrhea for ≥ 12 months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH and estradiol in the post-menopausal range per local standards.
  * If a patient is taking tamoxifen or toremifene and is aged < 60, then FSH and plasma estradiol levels should be in post-menopausal range per local values.
  * For women with therapy-induced amenorrhea, measurement of FSH and/or estradiol are needed to ensure menopausal status.
* Life expectancy ≥ 12 weeks.
* Locally advanced or metastatic breast cancer not amenable to curative intent.
* Histologically confirmed HR-positive/HER2-negative disease based on the most recent biopsy before signing the informed consent.

  * HER2 negativity is defined as either of the following by local laboratory assessment: IHC 0, IHC 1+ or IHC2+/in situ hybridisation (ISH/FISH) negative as per American Society of Clinical Oncology (ASCO)-College of American Pathologists Guideline (CAP) guideline(73).
  * ER and/or PR positivity are defined as >1% of cells expressing HR via IHC analysis as per ASCO-CAP guideline (74)
* Patients must have a site of disease amenable to safely perform a biopsy, as per Investigator's assessment, and be a candidate for tumor biopsy according to the treating institution's guidelines.
* Possibility of performing a biopsy prior to the start of treatment and its repetition after 2 weeks (14-21 days) on the same location. It will be provided formalin-fixed paraffin-embedded (FFPE) tumor block. The tumor tissue should be of good quality based on total and viable tumor content and must be evaluated centrally for PAM50 analysis prior to enrollment. Patients whose tumor tissue is not evaluable for central testing are not eligible. It is recommended to send the biopsy directly to the central lab after confirming the existence of a tumor, so as not to delay the inclusion, without the need to carry out IHC studies in the same.

  * Acceptable samples include core needle biopsies for deep tumor tissue or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions or biopsies from bone metastases.
  * Fine needle aspiration, brushing, cell pellet from pleural effusion and lavage samples are not acceptable.
* Patient must be willing to provide biopsy prior to the start of treatment and its repetition after 2 weeks (14-21 days) on the same location.
* The following subtypes identified in the pre-treatment tumor biopsy, as assessed by PAM50 assay at the Central Laboratory:

  * HER2-E (Cohort A)
  * Luminal A and Luminal B (Cohort B).
* No more than 4 prior lines of chemotherapy regimens for recurrent, locally advanced or metastatic breast cancer.
* Endocrine resistant disease, defined as the presence of disease recurrence while receiving adjuvant endocrine therapy for early stage breast cancer or disease progression of locally advanced/metastatic BC under ongoing endocrine therapy. There is no limit of previous received hormonal agents.
* Measurable and non-measurable (but evaluable) disease per RECIST 1.1 criteria.
* Adequate organ function, as determined by the following laboratory tests, within 28 days prior to enrollment:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  * Hemoglobin (Hb) ≥ 9 g/dL (red blood cell transfusion and/or erythropoietin allowed 7 days before study treatment).
  * Platelets ≥ 75,000/mm3.
  * International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) within therapeutic range
  * Serum creatinine ≤ 1.5x upper limit of normal (ULN)
  * AST or ALT ≤ 3 x ULN.
  * Serum bilirubin ≤ 1.5 upper limit of normal (ULN) unless the patient has documented non-malignant disease (e.g. Gilbert´s syndrome).
* Ability to swallow study drug and comply with study requirements.
* Resolution of all acute toxic effects of prior therapy or surgical procedures to baseline or Grade ≤ 1 (except alopecia or other toxicities not considered to be a safety risk for the patient) according to NCI CTCAE version 5.0.

Exclusion Criteria:

* History of current or previously treated CNS metastases or leptomeningeal disease. Testing for CNS metastasis is not mandatory.
* History of seizure or any condition that may predispose to seizure.
* Clinically significant cardiovascular disease within 6 months prior to enrolment defined as:

  * Myocardial infarction.
  * Inadequately controlled angina or serious cardiac arrhythmia not controlled by adequate medication.
  * Congestive heart failure (CHF) New York Health Association (NYHA) Class ≥ II.
  * History of clinically significant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, torsade de pointes).
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place.
  * Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) on 2 consecutive measurements at the screening visit.
  * Bradycardia as indicated by a heart rate of < 50 beats per minute on the screening electrocardiogram (ECG) recording.
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg on 2 consecutive measurements at the screening visit.
* Inability to swallow tablets, extensive reduction surgery of the stomach or small bowel or any active gastrointestinal disorder which may impair the absorption of the trial treatment (e.g. active peptic ulcer disease; uncontrolled celiac disease).
* Major surgical procedure within 4 weeks prior to allocation or anticipation of the need for major surgery during the course of study treatment.
* Use of medications that could reduce seizure threshold or concomitant treatment with potent CYP3A4 inducers.
* Treatment with warfarin and coumarin-like anticoagulants. Prophylactic use of low molecular weight heparin (LMWH) is allowed.
* Fructose intolerance.
* Treatment with any anticancer commercially available or investigational drug within 14 days prior to commencing trial treatment.
* Hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene.
* Current severe disease, infection, or systemic condition that renders the patient inappropriate for enrollment in the opinion of the investigator.
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of enzalutamide.
* Treatment with any approved or investigational agent that blocks androgen synthesis or targets the AR (eg, abiraterone acetate, ARN-509, bicalutamide, enzalutamide, ODM-201, TAK-448, TAK-683, TAK-700); or patients who progressed on Exemestane in adjuvant/advanced setting are not allowed; patients who received treatment for < 28 days or placebo on an investigational study are acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
changes of the PAM50 11-gene proliferation signature | after 2 weeks (14-21 days) of treatment with enzalutamide
  Relative changes of the PAM50 11-gene proliferation signature after 2 weeks (14-21 days) of treatment with enzalutamide. These changes will be analyzed according to the formula: Mean suppression = 100 - [geometric mean (post-treatment / pretreatment · 100)].

SECONDARY OUTCOMES:
Incidence, duration and severity of Adverse Events | during and after 2 weeks (14-21 days) of treatment with enzalutamide
  Incidence, duration and severity of Adverse Events (AEs) assessed by the NCI Common Terminology for Classification of Adverse Events (CTCAE) version 5, including dose reductions, delays and treatment discontinuations.
Relative changes of 33 gene signatures | after 2 weeks (14-21 days) of treatment with enzalutamide
  Relative changes of 33 gene signatures and 770 genes after 2 weeks (14-21 days) of treatment with enzalutamide and from week 3 to progression (in those patients who consent for optional biopsy). This study will be performed using the nCounter Breast 360TM panel.
  Relative changes of 33 gene signatures and 770 genes after 2 weeks (14-21 days) of treatment with enzalutamide and from week 3 to progression (in those patients who consent for optional biopsy). This study will be performed using the nCounter Breast 360TM panel.
somatic mutations | after 2 weeks (14-21 days) of treatment with enzalutamide
  Proportion of somatic mutations in samples from both cohorts using a targeted gene sequencing panel.
AR expression by IHC | before and after 21 days of treatment in Cohorts A and B.
  Analysis of AR expression by IHC (% nuclear expression in tumoral cell)
changes in percentage of cells expressing Ki67 by IHC | after 21 days of enzalutamide in HER2-E and Luminal A/B tumors.
  Relative changes in percentage of cells expressing Ki67
changes of It-TIL and Str-TIL | pre- and after 2 weeks (14-21 days) of treatment with enzalutamide and progression
  Analysis of lymphocyte infiltrate on hematoxylin and eosin-stained FFPE-sections. Percentage (%) change in It-TILs and Str-TILs infiltration
ctDNA levels | during and after 2 weeks (14-21 days) of treatment with enzalutamide
  Quantification of baseline ctDNA levels and 2 weeks (14-21 days) post-treatment. Determination of quantitative changes at day 21, at progression or at the end of trial due to other reasons
tumor ORR | after 2 weeks (14-21 days) of treatment with enzalutamide
  Proportion of patients who have a partial (PR) or complete response (CR) to therapy.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - ICO Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d' Hebrón, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación de Alcorcón, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No